CLINICAL TRIAL: NCT04608864
Title: Varicocele Repair for Infertile Men Undergoing IVF/ICSI: a Parallel, Two-group, Randomized Trial
Brief Title: Varicocele Repair for Men Undergoing IVF/ICSI
Acronym: Varicocele
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Yasmeen Fertility and Gynecology Center (Other)
Collaborators: Elite Fertility and Gynecology Center, Cairo, Egypt (Unknown); Banon IVF Center Assiut, Egypt (Other); IbnSina IVF Center, Sohag, Egypt (Unknown); Qena IVF Centre, Qena, Egypt (Unknown); Amshaj IVF Center (Other)
Responsible Party: Principal Investigator, Yasmin Magdi, Principal Investigator, Al-Yasmeen Fertility and Gynecology Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 008-2020
Record Dates: First submitted 2020-10-11; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- varicocelectomy arm (Experimental): The varicocelectomy procedure will be performed three months before ICSI for men with with male-factor infertility and were diagnosed clinically with varicocele
  Interventions: Procedure: varicocelectomy
- Control (No varicocelectomy) arm (No Intervention): Couples with male-factor infertility and males were diagnosed clinically with varicocele will undergo ICSI

INTERVENTIONS:
Procedure: varicocelectomy — microsurgical subinguinal varicocelectomy
  Other Names: varicocele repair
  Arms: varicocelectomy arm

SUMMARY:
For infertile men undergoing intracytoplasmic sperm injection (ICSI), data from retrospective studies suggested that varicocele repair may be beneficial and associated with improved livebirth and pregnancy rates, however, its role remains uncertain and disputed. To date, the investigators are not aware of published randomized controlled trail (RCT) that have evaluated whether varicocele repair would improve ICSI outcomes on patients with male-factor infertility.

DETAILED DESCRIPTION:
Varicocele repair in the era of assisted reproductive technology (ART) has been a point of dispute. The American Society for Reproductive Medicine (ASRM) Practice Committee recommended has considered ART as a primary treatment for female factor, regardless of the presence of varicocele and abnormal semen parameters.

A systematic review of 7 studies involving 1,241 men with a clinical varicocele and abnormal semen parameters showed improved livebirth and pregnancy rates after varicocelectomy in infertile men undergoing IVF/ICSI. Studies included in this systematic review were retrospective nature with a considerable heterogeneity. Evidence to support varicocelectomy for men with abnormal semen analysis undergoing IVF/ICSI has therefore remained inconclusive.

ELIGIBILITY:
Inclusion Criteria:

1. Couples able to provide informed consent.
2. Couples with at least 12 months of infertility
3. Couples with male-factor infertility
4. Couples counseled for ICSI procedure by reproductive specialist.
5. Couples undergoing their first ICSI cycle or their second ICSI cycle after a previously successful treatment.
6. Female: age between 18-43; body mass index (BMI) between 19.0-35.0 kg/m2; FSH level 3.0-20.0 miU/mL and/or AMH ≥1.5 pmol/L; with regular menstrual cycles (defined as 25 to 35 days in duration), evidence of ovulation (by biphasic basal body temperature, ovulation predictor kits, or luteal serum progesterone level ≥3 ng/mL), have no uterine abnormality by ultrasound; anticipated normal responder (≥5 antral follicle count or ≥5.4 pmol/L Anti- mullerian hormone (AMH).
7. Male: age: 18-55; able to produce freshly ejaculated sperm for the treatment cycle; diagnosed with clearly palpable varicocele; have at least one abnormal semen parameter on a semen analysis in the preceding 3 months: sperm concentration ≤15 million/mL (oligospermia), total motility≤40% (asthenospermia), or normal morphology ≤4% (teratospermia); normal hormonal profile

Exclusion Criteria:

1. Patients who willing to undergo ICSI with preimplantation genetic diagnosis.
2. Female: have previous two cycles of implantation failure at fresh transfer; with unilateral oophorectomy; PCOs; have any uterine pathology (myomas, adenomyosis, endocrinopathies, thrombophilia, chronic pathologies, acquired or congenital uterine abnormalities); have severe endometriosis; have uni- or bilateral hydrosalpinx; have history of recurrent pregnancy loss, takes any medical condition that affect fertility.
3. Male: have varicocele associated with hydrocele or inguinal hernia; secondary and recurrent varicocele, varicocele complicated by thrombophlebitis; varicocele with infertility due to other causes (demonstrated by andrologists), if they have a sperm concentration <1 million/mL on the screening semen analysis or if they were taking fertility medication or testosterone. Men are required to refrain from taking any medications for 4 weeks before randomization.
4. Abnormal karyotyping for female or male partners.
5. Uncontrolled diabetes, liver or renal disease, history of malignancy or borderline pathology of male or female partners.
6. Previous participation in the trial.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 2000 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Livebirth rate | up to 37 weeks
  the percentage of women who underwent randomization and will have a livebirth after at least 37 completed weeks of gestation

SECONDARY OUTCOMES:
Biochemical pregnancy | up to 2 weeks
  positive βhCG ≥10 IU/L at 14 days after egg retrieval
Clinical pregnancy | up to 7 weeks
  registered sacs with a heartbeat on ultrasound >7th week of gestation
Ongoing pregnancy | up to 20 weeks
Miscarriage | up to 20th weeks
stillbirth | up to 20 weeks
  intrauterine death at >20 weeks
Fertilization rate | up to 16-18 hours after ICSI
  number of oocytes fertilized per oocytes retrieved
Top quality embryos | up to 3 days after ICSI
  number of top quality embryos at Day 3 per number of fertilized oocytes
cryopreservation rate | up to 3-6 days after ICSI
  number of embryos cryopreserved per randomized woman
Blastocyst formation rate | up to 5 or 6 days after ICSI
  number of blastocyst at Day 5 or 6 per number of fertilized oocytes
implantation rate | up to 7 weeks
  number of intrauterine gestational sacs detected by ultrasound over the total number of embryos transferred

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Fawzy, Ph.D, Study Director — IbnSina IVF Center, IbnSina Hospital, Sohag

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3-6 months

REFERENCES:
- [Result] Kohn TP, Kohn JR, Pastuszak AW. Varicocelectomy before assisted reproductive technology: are outcomes improved? Fertil Steril. 2017 Sep;108(3):385-391. doi: 10.1016/j.fertnstert.2017.06.033. PMID 28865536
- [Result] Kirby EW, Wiener LE, Rajanahally S, Crowell K, Coward RM. Undergoing varicocele repair before assisted reproduction improves pregnancy rate and live birth rate in azoospermic and oligospermic men with a varicocele: a systematic review and meta-analysis. Fertil Steril. 2016 Nov;106(6):1338-1343. doi: 10.1016/j.fertnstert.2016.07.1093. Epub 2016 Aug 12. PMID 27526630
- [Result] Practice Committee of the American Society for Reproductive Medicine; Society for Male Reproduction and Urology. Report on varicocele and infertility: a committee opinion. Fertil Steril. 2014 Dec;102(6):1556-60. doi: 10.1016/j.fertnstert.2014.10.007. Epub 2014 Nov 25. PMID 25458620